CLINICAL TRIAL: NCT03822117
Title: A Phase 2, Open-Label, Single-Arm, Multicenter Study to Evaluate the Efficacy and Safety of Pemigatinib in Participants With Previously Treated Locally Advanced/Metastatic or Surgically Unresectable Solid Tumor Malignancies Harboring Activating FGFR Mutations or Translocations (FIGHT-207)
Brief Title: Efficacy and Safety of Pemigatinib in Previously Treated Locally Advanced/Metastatic or Surgically Unresectable Solid Tumor Malignancies Harboring Activating FGFR Mutations or Translocations (FIGHT-207)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A business decision was made to to discontinue further enrollment. There were no safety concerns that contributed to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-207; 2018-004768-69 (EudraCT Number)
Expanded Access: NCT03906357 (No longer available)
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Results first posted 2023-03-15 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor Malignancy
Keywords: Fibroblast growth factor receptor (FGFR) inhibitor; FGFR mutations; FGFR translocations; solid tumor malignancy
MeSH Terms: conditions — Acrocephalosyndactylia | interventions — pemigatinib

STUDY DESIGN:
Intervention Model Description: This study consists of 3 cohorts that will have study drug administered in parallel, Cohort A, Cohort B, and Cohort C. There is no difference in the treatment regimen between the cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pemigatinib (Experimental): Cohort A (Solid tumor malignancies with FGFR1-3 in frame fusions; any FGFR2 rearrangement; FGFR1/3 rearrangement with known partner*). Cohort B (Solid tumor malignancies with known or likely activating mutations (excluding kinase domain) in FGFR1-3) Cohort C (Solid tumor malignancies with FGFR1-3 known activating mutations in kinase domain; FGFR1-3 putatively activating mutations; other FGFR1/3 rearrangements* (not eligible for Cohort A)).
  *Only FGFR fusions or rearrangements with an intact kinase domain are eligible
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib administered orally once daily (QD).
  Other Names: INCB054828

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pemigatinib in participants with previously treated locally advanced/metastatic or surgically unresectable solid tumor malignancies harboring activating FGFR mutations or translocations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor malignancy that is advanced or metastatic or is surgically unresectable.
* Radiographically measurable disease (per RECIST v1.1 or RANO for primary brain tumors). Tumor lesions located in a previously irradiated area or in an area subjected to other loco-regional therapy are considered measureable if progression has been clearly demonstrated in the lesion.
* Documentation of an FGFR1-3 gene mutation or translocation.
* Objective progression after at least 1 prior therapy and no therapy available that is likely to provide clinical benefit. Participants who are intolerant to or decline the approved therapy are eligible only if they have no therapy available that is likely to provide clinical benefit.
* Eastern Cooperative Oncology Group performance status 0 to 2.
* Baseline archival tumor specimen (if less than 24 months from date of screening) or willingness to undergo a pretreatment tumor biopsy to obtain the specimen. Must be a tumor block or approximately 15 unstained slides from biopsy or resection of primary tumor or metastasis.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Prior receipt of a selective FGFR inhibitor in the past 6 months.
* Receipt of anticancer medications or investigational drugs for any indication or reason within 28 days before first dose of pemigatinib.
* Cannot be a candidate for potentially curative surgery.
* Current evidence of clinically significant corneal or retinal disorder as confirmed by ophthalmologic examination.
* Radiation therapy administered within 2 weeks of enrollment/first dose of study treatment.
* Untreated brain or central nervous system (CNS) metastases or brain or CNS metastases that have progressed (eg, evidence of new or enlarging brain metastasis or new neurological symptoms attributable to brain or CNS metastases).
* Known additional malignancy that is progressing or requires active treatment.
* History of calcium and phosphate hemostasis disorder or systemic mineral imbalance with ectopic calcification of soft tissues.
* Clinically significant or uncontrolled cardiac disease.
* Active chronic or current infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment within 2 weeks before enrollment (participants with asymptomatic chronic infections on prophylactic treatment are allowed).
* Evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (defined as elevated transaminases or cirrhosis; chronic HBV/HCV infection with no cirrhosis and no elevated transaminases is allowed).
* Known HIV infection.
* Use of any potent CYP3A4 inhibitors or inducers or moderate CYP3A4 inducers within 14 days or five half-lives (whichever is longer) before the first dose of study drug/treatment.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — Incyte Corporation
Locations (90):
- United States (44):
  - Cancer Treatment Centers of America, Goodyear, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Chao Family Comprehensive Cancer Center University of California, Irvine, Orange, California
  - Stanford Cancer Center, Palo Alto, California
  - John Wayne Cancer Institute, Santa Monica, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Florida Cancer Specialists & Research Institute, Fort Myers, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Edward H Kaplan & Associates, Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Cancer Treatment Centers of America, Zion, Illinois
  - Indiana University Health - Arnett Cancer Care, Lafayette, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Ochsner Clinic, New Orleans, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Umass Memorial Medical Center, Inc., Worcester, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Summit Medical Group, Florham Park, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Southwestern Regional Medical Center, Tulsa, Oklahoma
  - Cancer Institute of Greenville Health System, Greenville, South Carolina
  - The West Clinic Pc, Germantown, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Joe Arrington Cancer Center, Lubbock, Texas
  - Virginia Cancer Specialists, Pc, Fairfax, Virginia
  - Virginia Oncology Associates-Lake Wright, Norfolk, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Multicare Institute For Research & Innovation, Tacoma, Washington
  - West Virginia University Hospitals Inc, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- The Finsen Centre National Hospital, Copenhagen, Denmark
- France (6):
  - Institut Bergonie, Bordeaux
  - CENTRE GEORGES FRANï¿½OIS LECLERC, Dijon
  - Centre Antoine Lacassagne, Nice
  - Hospital Saint Louis, Paris
  - A.P.H. Paris Hopital Cochin, Paris
  - Institut Universitaire Du Cancer de Toulouse Oncopole, Toulouse
- Germany (5):
  - Universitatsklinikum Koln, Cologne
  - University Medical Center Freiburg, Freiburg im Breisgau
  - University Medical Centre Hamburg-Eppendorf, Centre of Oncology, Hamburg
  - University Hospital Grosshadern Munich, Munich
  - Universitaetsklinikum in Tubingen, Tübingen
- Israel (5):
  - Ha Emek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - Hadassah Hebrew University Medical Center Ein Karem Hadassah, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (6):
  - L AZIENDA OSPEDALIERO-UNIVERSITARIA DI BOLOGNA POLICLINICO S. ORSOLA ï¿½ MALPIGHI, Bologna
  - Fondazione Del Piemonte Per L Oncologia Ircc Candiolo, Candiolo
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Napoli
  - Istituto Nazionale Tumori Regina Elena Irccs, Roma
  - Centro Ricerche Cliniche Di Verona (Crc), Verona
- Japan (7):
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kanazawa University Hospital, Ishikawa
  - Kobe University Hospital, Kobe
  - Tohoku University Hospital, Sendai
  - Keio University Hospital, Shinjuku-ku
  - Shizuoka Cancer Center, Shizuoka
  - Kanagawa Cancer Center, Yokohama
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Centro Integral Oncologico Clara Campal (Ciocc), Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinica Universidad de Navarra (Cun), Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Y Politcnico de La Fe, Valencia
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Universitatsspital Zurich, Zurich
- United Kingdom (3):
  - University College London Hospitals (Uclh), London
  - Imperial College Healthcare Nhs Trust - Hammersmith Hospital, London
  - Sarah Cannon Research Institute, London

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Rodon J, Damian S, Furqan M, Garcia-Donas J, Imai H, Italiano A, Spanggaard I, Ueno M, Yokota T, Veronese ML, Oliveira N, Li X, Gilmartin A, Schaffer M, Goyal L. Pemigatinib in previously treated solid tumors with activating FGFR1-FGFR3 alterations: phase 2 FIGHT-207 basket trial. Nat Med. 2024 Jun;30(6):1645-1654. doi: 10.1038/s41591-024-02934-7. Epub 2024 May 6. PMID 38710951

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study enrolled participants at 49 study sites in the United States, South Korea, United Kingdom, France, Italy, Israel, Germany, Spain, Denmark, and Japan.
Groups:
- Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements: Participants with fibroblast growth factor receptor (FGFR) 1-3 in-frame fusions or fibroblast growth factor receptor 2 (FGFR2) rearrangements self-administered oral pemigatinib at a starting dose of 13.5 milligrams (mg) once daily (QD) continuously in 21-day cycles. Pemigatinib was administered until documented disease progression or unacceptable toxicity.
- Cohort B: Known or Likely Activating FGFR1-3 Mutations: Participants with known or likely activating mutations in FGFR1-3 self-administered oral pemigatinib at a starting dose of 13.5 mg QD continuously in 21-day cycles. Pemigatinib was administered until documented disease progression or unacceptable toxicity.
- Cohort C: Other FGFR Mutations or Arrangements: Participants with other FGFR mutations or arrangements self-administered oral pemigatinib at a starting dose of 13.5 mg QD continuously in 21-day cycles. Pemigatinib was administered until documented disease progression or unacceptable toxicity.
- Other: Participants with an FGF/FGFR status for whom the local laboratory FGF/FGFR results could not be confirmed centrally self-administered oral pemigatinib at a starting dose of 13.5 mg QD continuously in 21-day cycles. Pemigatinib was administered until documented disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements | Cohort B: Known or Likely Activating FGFR1-3 Mutations | Cohort C: Other FGFR Mutations or Arrangements | Other
Started | 49 | 32 | 26 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 49 | 32 | 26 | 4
Not completed — Death | 18 | 17 | 12 | 4
Not completed — Lost to Follow-up | 1 | 2 | 3 | 0
Not completed — Study Terminated by Sponsor | 25 | 11 | 6 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 3 | 0
Not completed — Disease Progression | 1 | 2 | 1 | 0
Not completed — Never Returned to Hospital | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements | Cohort B: Known or Likely Activating FGFR1-3 Mutations | Cohort C: Other FGFR Mutations or Arrangements | Other | Total
Number analyzed (Participants) | 49 | 32 | 26 | 4 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (11.51) | 66.0 (10.04) | 61.5 (13.32) | 48.0 (14.45) | 61.4 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 19 | 14 | 1 | 62
  Male | 21 | 13 | 12 | 3 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 38 | 20 | 16 | 0 | 74
  Black or African American | 0 | 0 | 1 | 0 | 1
  Asian | 9 | 9 | 7 | 4 | 29
  Participant Declined to Provide | 1 | 0 | 0 | 0 | 1
  Not Available | 0 | 1 | 0 | 0 | 1
  Not Required in Country of Origin | 0 | 1 | 0 | 0 | 1
  Missing | 1 | 1 | 2 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 44 | 25 | 20 | 3 | 92
  Not Reported | 2 | 2 | 3 | 1 | 8
  Unknown | 1 | 2 | 0 | 0 | 3
  Captured as "Other" | 0 | 1 | 0 | 0 | 1
  Missing | 1 | 1 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), Defined as the Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR) Based on RECIST v1.1 or RANO, in Participants With FGFR1-3 In-frame Fusions or FGFR2 Arrangements
Description: Per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1): CR: disappearance of all target/non-target lesions; no appearance of new lesions. PR: complete disappearance or a ≥30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters; no new lesions; no progression of non-target lesions. Per Response Assessment in Neuro-Oncology (RANO; for participants with primary brain tumors): CR: disappearance of all enhancing lesions; stable/improved non-enhancing lesions; stable/improved clinically. PR: ≥50% decrease in sum of perpendicular diameters of measurable enhancing lesions; no progression of non-measurable disease; stable/improved non-enhancing lesions; stable/improved clinically. Cohort determination was based on FGFR status from a central genomics laboratory. Response data were from an independent centralized radiological review committee per RECIST v1.1 and RANO, and response was confirmed.
Time Frame: up to 483 days
Population: Efficacy Evaluable Population: all enrolled participants in Cohorts A, B, and C who received at least 1 dose of pemigatinib. Confidence interval was calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements | Cohort B: Known or Likely Activating FGFR1-3 Mutations | Cohort C: Other FGFR Mutations or Arrangements | Other
Number analyzed (Participants) | 49 | 0 | 0 | 0
percentage of participants | 26.5 [14.95 to 41.08] |  |  |

2. Primary Outcome: ORR, Defined as the Percentage of Participants With a Best Overall Response of CR or PR Based on RECIST v1.1 or RANO, in Participants With Known or Likely Activating FGFR1-3 Mutations
Description: Per RECIST v1.1: CR: disappearance of all target/non-target lesions; no appearance of new lesions. PR: complete disappearance or a ≥30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters; no new lesions; no progression of non-target lesions. Per RANO (for participants with primary brain tumors): CR: disappearance of all enhancing lesions; stable/improved non-enhancing lesions; stable/improved clinically. PR: ≥50% decrease in sum of perpendicular diameters of measurable enhancing lesions; no progression of non-measurable disease; stable/improved non-enhancing lesions; stable/improved clinically. Cohort determination was based on FGFR status from a central genomics laboratory. Response data were from an independent centralized radiological review committee per RECIST v1.1 and RANO, and response was confirmed.
Time Frame: up to 449 days
Population: Efficacy Evaluable Population. Confidence interval was calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements | Cohort B: Known or Likely Activating FGFR1-3 Mutations | Cohort C: Other FGFR Mutations or Arrangements | Other
Number analyzed (Participants) | 0 | 32 | 0 | 0
percentage of participants |  | 9.4 [1.98 to 25.02] |  |

3. Secondary Outcome: Progression-free Survival (PFS) in Participants With FGFR1-3 In-frame Fusions or FGFR2 Arrangements and in Participants With Known or Likely Activating FGFR1-3 Mutations
Description: PFS was defined as the time from the first dose until progressive disease (according to RECIST v1.1 or RANO for participants with primary brain tumors and assessed by an independent centralized radiological review committee) or death (whichever occurred first).
Time Frame: up to 532 days
Population: Efficacy Evaluable Population. The 95% confidence interval is calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements | Cohort B: Known or Likely Activating FGFR1-3 Mutations | Cohort C: Other FGFR Mutations or Arrangements | Other
Number analyzed (Participants) | 49 | 32 | 0 | 0
months | 4.53 [3.58 to 6.28] | 3.68 [2.07 to 4.47] |  |

4. Secondary Outcome: Duration of Response (DOR), Defined as the First CR or PR Assessment Until Progressive Disease (PD) or Death, in Participants With FGFR1-3 In-frame Fusions or FGFR2 Arrangements and in Participants With Known or Likely Activating FGFR1-3 Mutations
Description: Assessment was by an independent centralized radiological review committee; response was confirmed. Per RECIST v1.1: CR: disappearance of all target (TLs)/non-target lesions (NTLs); no appearance of new lesions. PR: complete disappearance or a ≥30% decrease in the sum of the diameters of TLs, taking as a reference the baseline sum diameters; no new lesions; no progression of NTLs. PD: progression of a TL/NTL or presence of new lesion. Per RANO (participants with primary brain tumors): CR: disappearance of all enhancing lesions (ELs); stable/improved non-enhancing lesions (NELs); stable/improved clinically. PR: ≥50% decrease in sum of perpendicular diameters of measurable ELs; no progression of non-measurable disease; stable/improved NELs; stable/improved clinically. PD: >25% increase in sum of perpendicular diameters of all measurable ELs; significant increase of NELs; new lesions; clear clinical deterioration; failure to return for evaluation due to death/deteriorating condition.
Time Frame: up to 24.90 months
Population: Efficacy Evaluable Population. The 95% confidence interval is calculated using the Brookmeyer and Crowley's method. Only participants with a CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements | Cohort B: Known or Likely Activating FGFR1-3 Mutations | Cohort C: Other FGFR Mutations or Arrangements | Other
Number analyzed (Participants) | 13 | 3 | 0 | 0
months | 7.79 [4.17 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 6.93 [4.01 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. |  |

5. Secondary Outcome: Overall Survival in Participants With FGFR1-3 In-frame Fusions or FGFR2 Arrangements and in Participants With Known or Likely Activating FGFR1-3 Mutations
Description: Overall survival was defined as the time from the first dose of study drug to death of any cause.
Time Frame: up to 532 days
Population: Efficacy Evaluable Population. The 95% confidence interval was calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements | Cohort B: Known or Likely Activating FGFR1-3 Mutations | Cohort C: Other FGFR Mutations or Arrangements | Other
Number analyzed (Participants) | 49 | 32 | 0 | 0
months | 17.48 [7.79 to NA] — The upper limit of the confidence interval was not estimable because too few participants had died. | 11.37 [6.57 to NA] — The upper limit of the confidence interval was not estimable because too few participants had died. |  |

6. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) and Any Treatment-related Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. TEAEs were defined as AEs reported for the first time or the worsening of pre-existing events after the first dose of study treatment. Treatment-related AEs were defined as TEAEs judged as related by the investigator or with a missing causality.
Time Frame: up to 651 days
Population: Safety Population: all enrolled participants who received at least 1 dose of pemigatinib
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements | Cohort B: Known or Likely Activating FGFR1-3 Mutations | Cohort C: Other FGFR Mutations or Arrangements | Other
Number analyzed (Participants) | 49 | 32 | 26 | 4
Participants
  TEAEs | 49 | 32 | 26 | 4
  Treatment-related AEs | 46 | 32 | 26 | 4

ADVERSE EVENTS:
Time Frame: up to 651 days
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events reported for the first time or the worsening of pre-existing events after the first dose of study treatment, are reported.
Groups:
- Total: Total
Arm/Group | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements | Cohort B: Known or Likely Activating FGFR1-3 Mutations | Cohort C: Other FGFR Mutations or Arrangements | Other | Total
All-Cause Mortality (participants affected / at risk) | 18/49 | 17/32 | 13/26 | 4/4 | 52/111
Serious Adverse Events (participants affected / at risk) | 21/49 | 7/32 | 10/26 | 2/4 | 40/111
Other Adverse Events (participants affected / at risk) | 49/49 | 32/32 | 26/26 | 4/4 | 111/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements (N=49) | Cohort B: Known or Likely Activating FGFR1-3 Mutations (N=32) | Cohort C: Other FGFR Mutations or Arrangements (N=26) | Other (N=4) | Total (N=111)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal erosion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cutaneous calcification (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fascial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Long QT syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stent malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: FGFR1-3 In-frame Fusions or FGFR2 Arrangements (N=49) | Cohort B: Known or Likely Activating FGFR1-3 Mutations (N=32) | Cohort C: Other FGFR Mutations or Arrangements (N=26) | Other (N=4) | Total (N=111)
Abdominal pain (Gastrointestinal disorders) | 7 (10) | 3 (3) | 5 (5) | 0 (0) | 15 (18)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (2) | 3 (3) | 0 (0) | 7 (8)
Agitation (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 6 (8) | 5 (5) | 3 (3) | 0 (0) | 14 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (20) | 17 (21) | 8 (8) | 0 (0) | 45 (49)
Anaemia (Blood and lymphatic system disorders) | 8 (9) | 4 (4) | 2 (2) | 0 (0) | 14 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (12) | 11 (14) | 1 (1) | 0 (0) | 23 (27)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 5 (9) | 4 (5) | 5 (6) | 0 (0) | 14 (20)
Asthenia (General disorders) | 8 (8) | 11 (15) | 8 (9) | 0 (0) | 27 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 8 (8)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Blood creatinine increased (Investigations) | 10 (10) | 3 (3) | 5 (5) | 0 (0) | 18 (18)
COVID-19 (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 2 (5)
Conjunctivitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 7 (8)
Constipation (Gastrointestinal disorders) | 18 (20) | 13 (18) | 6 (6) | 0 (0) | 37 (44)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7) | 2 (2) | 0 (0) | 11 (12)
Cystitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 10 (14) | 12 (15) | 5 (5) | 0 (0) | 27 (34)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 19 (28) | 17 (30) | 7 (7) | 0 (0) | 43 (65)
Dizziness (Nervous system disorders) | 5 (5) | 1 (3) | 1 (1) | 0 (0) | 7 (9)
Dry eye (Eye disorders) | 12 (13) | 9 (10) | 4 (5) | 0 (0) | 25 (28)
Dry mouth (Gastrointestinal disorders) | 13 (15) | 11 (13) | 7 (8) | 1 (1) | 32 (37)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7) | 6 (7) | 5 (6) | 1 (1) | 18 (21)
Dysgeusia (Nervous system disorders) | 10 (12) | 14 (17) | 6 (7) | 0 (0) | 30 (36)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5) | 2 (2) | 0 (0) | 9 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 9 (9)
Erythema (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Fatigue (General disorders) | 10 (14) | 9 (11) | 4 (4) | 0 (0) | 23 (29)
Headache (Nervous system disorders) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 7 (7)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (4) | 3 (3) | 3 (8) | 0 (0) | 8 (15)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 45 (72) | 27 (51) | 17 (27) | 4 (4) | 93 (154)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (2) | 0 (0) | 1 (1) | 7 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 6 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 2 (4) | 1 (1) | 10 (12)
Hypotension (Vascular disorders) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 6 (8)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Keratitis (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Lipase increased (Investigations) | 2 (3) | 1 (1) | 2 (3) | 0 (0) | 5 (7)
Malaise (General disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 4 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 10 (10)
Nail discolouration (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4) | 2 (2) | 0 (0) | 13 (13)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 2 (2) | 0 (0) | 10 (10)
Nail infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 11 (12) | 8 (12) | 6 (7) | 2 (2) | 27 (33)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 6 (6) | 5 (5) | 2 (2) | 0 (0) | 13 (13)
Onychalgia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Onycholysis (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (6) | 3 (3) | 0 (0) | 10 (12)
Onychomadesis (Skin and subcutaneous tissue disorders) | 7 (8) | 6 (6) | 4 (4) | 0 (0) | 17 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 0 (0) | 3 (3) | 0 (0) | 10 (11)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 (15) | 8 (11) | 5 (5) | 0 (0) | 26 (31)
Paronychia (Infections and infestations) | 5 (5) | 6 (7) | 3 (3) | 0 (0) | 14 (15)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 6 (6)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 5 (5)
Serous retinal detachment (Eye disorders) | 5 (6) | 3 (3) | 1 (1) | 0 (0) | 9 (10)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 27 (39) | 17 (25) | 13 (21) | 2 (2) | 59 (87)
Taste disorder (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 4 (5)
Urinary retention (Renal and urinary disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 6 (6)
Urinary tract infection (Infections and infestations) | 6 (6) | 5 (5) | 4 (5) | 0 (0) | 15 (16)
Vision blurred (Eye disorders) | 5 (5) | 3 (4) | 0 (0) | 0 (0) | 8 (9)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 4 (5)
Vomiting (Gastrointestinal disorders) | 10 (14) | 5 (6) | 5 (5) | 0 (0) | 20 (25)
Weight decreased (Investigations) | 8 (9) | 6 (6) | 2 (2) | 0 (0) | 16 (17)
Xerosis (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03822117/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03822117/SAP_001.pdf